CLINICAL TRIAL: NCT04776018
Title: A Phase 1b/2 Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of TAK-981 in Combination With Monoclonal Antibodies in Adult Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study Of TAK-981 Given With Monoclonal Antibodies (mAbs) In Adults With Relapsed or Refractory Multiple Myeloma (RRMM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-981-1503
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma (RRMM)
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-981; daratumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Phase 1b, Part 1 - Dose Escalation: Arm A - TAK-981 Twice Weekly (BIW) + Mezagitamab (Experimental): Mezagitamab: A fixed dose of 600 mg subcutaneous (SC) injection once weekly in Cycles 1 and 2 (each cycle is of 28 days), followed by once every 2 weeks in Cycle 3 through 6, then every 4 weeks up to Cycle 24 or until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  TAK-981: Escalating doses of TAK-981 BIW intravenous (IV) infusion on Days 1, 4, 8, 11 and 15 in Cycle 1 and 2 (each Cycle is of 28 days) followed by every 2 weeks in Cycles 3 through 6, followed by once every 4 weeks up to Cycle 24 or until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  Interventions: Drug: TAK-981; Drug: Mezagitamab
- Phase 1b, Part 1 - Dose Escalation: Arm B - TAK-981 Weekly (QW) + Mezagitamab (Experimental): Mezagitamab: A fixed dose of 600 mg SC injection once weekly in Cycles 1 and 2 (each cycle is of 28 days), followed by once every 2 weeks from Cycle 3 through 6, then every 4 weeks up to Cycle 24 or until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  TAK-981: Escalating doses of TAK-981 QW IV infusion on Days 1, 8, 15, and 22 in Cycles 1 and 2 (each cycle is of 28 days), followed by every 2 weeks in Cycles 3 through 6, followed by once every 4 weeks. up to Cycle 24 or until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  Interventions: Drug: TAK-981; Drug: Mezagitamab
- Phase 1b, Part 2 - Lead-in Cohort: TAK-981 + Daratumumab and Hyaluronidase-fihj (Experimental): Daratumumab and hyaluronidase-fihj: 1800 mg SC injection QW once weekly in Cycles 1 and 2 , (each cycle is of 28 days) followed by every 2 weeks in Cycle 3 through 6 , followed by every 4 weeks up to Cycle 24 until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  TAK-981: As per dose and schedule of TAK-981 defined in Phase 1b Part 1.
  Interventions: Drug: TAK-981; Drug: Daratumumab and Hyaluronidase-fihj
- Phase 2 - Dose Expansion: TAK-981 + Daratumumab and Hyaluronidase-fihj or Mezagitamab (Experimental): TAK-981 at RP2D as determined in Phase 1b. Mezagitamab at a fixed dose of 600 mg SC injection or Daratumumab and Hyaluronidase-fihj at a fixed dose of 1800 mg weekly in Cycles 1 and 2 (each cycle is of 28 days), followed by every 2 weeks in Cycle 3 through 6, followed by every 4 weeks up to Cycle 24 or until disease progression unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  Interventions: Drug: TAK-981; Drug: Mezagitamab; Drug: Daratumumab and Hyaluronidase-fihj

INTERVENTIONS:
Drug: TAK-981 — TAK-981 IV infusion.
Drug: Mezagitamab — Mezagitamab SC injection.
  Arms: Phase 1b, Part 1 - Dose Escalation: Arm A - TAK-981 Twice Weekly (BIW) + Mezagitamab; Phase 1b, Part 1 - Dose Escalation: Arm B - TAK-981 Weekly (QW) + Mezagitamab; Phase 2 - Dose Expansion: TAK-981 + Daratumumab and Hyaluronidase-fihj or Mezagitamab
Drug: Daratumumab and Hyaluronidase-fihj — Daratumumab and Hyaluronidase-fihj SC injection.
  Arms: Phase 1b, Part 2 - Lead-in Cohort: TAK-981 + Daratumumab and Hyaluronidase-fihj; Phase 2 - Dose Expansion: TAK-981 + Daratumumab and Hyaluronidase-fihj or Mezagitamab

SUMMARY:
TAK-981 is being tested in combination with anti-CD38 monoclonal antibodies (mAbs) to treat participants who have relapsed or refractory multiple myeloma (RRMM).

The main aims of the study are to evaluate the safety and efficacy of TAK-981 in combination with anti-CD38 (mAbs) and to determine the recommended Phase 2 dose (RP2D).

Participants will be on this combination treatment for 28-day cycles. They will continue with this treatment until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-981. TAK-981 in combination with an anti-CD38 monoclonal antibody (mAbs) is being tested to treat people who have RRMM. The study will include a dose escalation phase and a dose expansion phase.

The study will enroll approximately 81 participants; approximately 30 participants in the dose escalation phase (Part 1) approximately 15 participants in (Part 2) and up to 36 participants in dose expansion phase (Part 2). Participants will receive escalating doses of TAK-981 in combination with fixed doses as follows:

* Phase 1b, Part 1 - Dose Escalation: Arm A - TAK-981 Twice Weekly (BIW) + Mezagitamab
* Phase 1b, Part 1 - Dose Escalation: Arm B - TAK-981 Weekly (QW) + Mezagitamab
* Phase 1b, Part 2 - Dose Escalation: TAK-981 + Daratumumab and Hyaluronidase-fihj

Once RP2D is determined in Phase 1, participants with RRMM will be enrolled in Phase 2.

• Phase 2 - Dose Expansion: TAK-981 + Daratumumab and Hyaluronidase-fihj or Mezagitamab

This multi-center trial will be conducted in North America. The overall time to participate in this study is 2 years. Participants will make multiple visits to the clinic, and progression-free survival follow-up for maximum up to 12 months after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have RRMM with measurable disease:

   a) Has measurable disease defined as one of the following:
   * Serum M-protein ≥0.5 g/dL (≥5 g/L).
   * Urine M-protein ≥200 mg/24 hours.
   * In participants without measurable M-protein in serum protein electrophoresis (SPEP) or urine protein electrophoresis (UPEP), a serum free light chain (FLC) assay result with involved FLC level ≥10 mg/dL (≥100 mg/L), provided serum FLC ratio is abnormal.
2. Has undergone stem cell transplant or is considered transplant ineligible.
3. Has failed at least 3 prior lines of anti-myeloma treatments and is either refractory, or intolerant to at least 1 immunomodulatory drug ( IMiD); (ie, lenalidomide or pomalidomide [thalidomide excluded]), at least 1 proteasome inhibitor (ie, bortezomib, ixazomib or carfilzomib), and refractory to at least 1 anti-CD38 antibody and who have demonstrated disease progression with the last therapy.

5.Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.

6.Have recovered to Grade 1 or baseline from all toxicity associated with previous therapy or have the toxicity established as sequela.

Exclusion Criteria:

1. Received treatment with systemic anticancer treatments within 14 days before the first dose of study drug.
2. Current participation in another interventional study, including other clinical trials with investigational agents (including investigational vaccines or investigational medical device for disease under study) within 4 weeks of the first dose of TAK-981 and throughout the duration of this trial.
3. Prior radiation therapy within 14 days of the first dose of TAK-981.
4. Major surgery within 4 weeks before C1D1. participants should be fully recovered from any surgically related complications.
5. Plasmapheresis within 28 days of randomization.
6. Diagnosis of primary amyloidosis, Waldenström's disease, monoclonal gammopathy of undetermined significance or smoldering multiple myeloma (SMM), plasma cell leukemia POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), myelodysplastic syndrome, or myeloproliferative syndrome.
7. With disease where the only measurable parameter is plasmacytoma.
8. Second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the participant is not on active anticancer therapy.
9. Prior treatment with more than 1 anti-CD38 antibody.
10. Requires the use of drugs known to prolong the corrected QT interval (QTc) (during Phase 1b only).
11. History of QT interval with Fridericia's correction (QTcF) >480 ms.
12. History of human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C infection.
13. Systemic infection requiring systemic antibiotic therapy.
14. Active or history pneumonitis.
15. Receipt of any live vaccine (eg, varicella, pneumococcus) within 4 weeks of initiation of study drug.
16. Receiving strong or moderate Cytochrome P450 (CYP) 3A4/5 inhibitors or inducers.
17. History of unstable cardiac comorbidities in the following 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (13):
- United States (12):
  - Mayo Clinic Arizona - PPDS, Scottsdale, Arizona
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Mayo Clinic - Cancer Center - Rochester - PPDS, Rochester, Minnesota
  - Oncology Hematology West (Omaha) - USOR, Omaha, Nebraska
  - Weill Cornell Medical Center, New York, New York
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - Baylor Sammons Cancer Center, Dallas, Texas
  - Northeast Texas Cancer and Research Institute, Tyler, Texas
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Nakamura A, Grossman S, Song K, Xega K, Zhang Y, Cvet D, Berger A, Shapiro G, Huszar D. The SUMOylation inhibitor subasumstat potentiates rituximab activity by IFN1-dependent macrophage and NK cell stimulation. Blood. 2022 May 5;139(18):2770-2781. doi: 10.1182/blood.2021014267. PMID 35226739
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/60423834eb9d7e001f5bc61b

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States and Canada from 20 April 2021 to 09 November 2023. Participants with diagnosis of Relapsed and/or Refractory Multiple Myeloma (RRMM) were enrolled in Phase 1b Part 1 to receive TAK-981 in combination with mezagitamab.
Pre-assignment Details: This study consisted of Phase 1b and 2. Phase 1b (Dose Escalation) had two parts (Parts 1 and 2) and Phase 2 (Dose Expansion) was single part. Phase 1b- Part 2 and Phase 2 were not conducted, as study was terminated early after completion of Phase 1b Part 1 due to business reasons and therefore, no data for Phase 1b Part 2 and Phase 2 was collected and reported.
Groups:
- Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg: Participants received TAK-981 60 milligrams (mg), infusion, intravenously, twice weekly (BIW) on Days 1, 4, 8, 11 and 15, and mezagitamab 600 mg, injection, subcutaneously, once weekly on Days 1, 8, 15 and 22 during Cycles 1 and 2, then once every 2 weeks during Cycles 3 through 6, further once every 4 weeks, until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg: Participants received TAK-981 90 mg, infusion, intravenously, twice weekly on Days 1, 4, 8, 11 and 15, and mezagitamab 600 mg, injection, subcutaneously, once weekly on Days 1, 8, 15 and 22 during Cycles 1 and 2, then once every 2 weeks during Cycles 3 through 6, further once every 4 weeks, until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg: Participants received TAK-981 90 mg, infusion, intravenously, in combination with mezagitamab 600 mg, injection, subcutaneously, once weekly (QW) on Days 1, 8, 15, 22 during Cycles 1 and 2, then every 2 weeks during Cycles 3 through 6, further once every 4 weeks until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg: Participants received TAK-981 120 mg, infusion, intravenously, twice weekly on Days 1, 4, 8, 11 and 15, and mezagitamab 600 mg, injection, subcutaneously, once weekly on Days 1, 8, 15 and 22 during Cycles 1 and 2, then once every 2 weeks during Cycles 3 through 6, further once every 4 weeks, until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg: Participants received TAK-981 120 mg, infusion, intravenously, in combination with mezagitamab 600 mg, injection, subcutaneously, once weekly on Days 1, 8, 15, 22 during Cycles 1 and 2, then every 2 weeks during Cycles 3 through 6, further once every 4 weeks until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Phase 1b, Part 2: TAK-981 + Daratumumab + Hyaluronidase-fihj: Participants were planned to receive TAK-981, infusion, intravenously, in combination with daratumumab and hyaluronidase-fihj, injection, subcutaneously, once weekly in Cycles 1 and 2, then every 2 weeks during Cycles 3 through 6, further once every 4 weeks until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days. No participants were enrolled in this arm as this study was terminated early before start of enrolment in Phase 1b, Part 2.
- Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody: Participants were planned to receive TAK-981 recommended phase 2 dose (RP2D), infusion, intravenously, in combination with an anti-CD38 antibody (mezagitamab or daratumumab and hyaluronidase-fihj), injection, subcutaneously, for up to 24 cycles or until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days. No participants were enrolled in this arm as this study was terminated early before start of enrolment in Phase 2.
Period: Overall Study
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg | Phase 1b, Part 2: TAK-981 + Daratumumab + Hyaluronidase-fihj | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Started | 3 | 3 | 10 | 3 | 8 | 0 (The study was terminated before start of enrolment in Phase 1b, Part 2. Hence, no participants were enrolled in Phase 1b Part 2.) | 0 (The study was terminated before start of enrolment in Phase 2. Hence, no participants were enrolled in Phase 2.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 10 | 3 | 8 | 0 | 0
Not completed — Death | 0 | 1 | 4 | 1 | 4 | 0 | 0
Not completed — Study terminated by sponsor | 2 | 1 | 4 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Groups:
- Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg: Participants received TAK-981 60 mg, infusion, intravenously, twice weekly on Days 1, 4, 8, 11 and 15, and mezagitamab 600 mg, injection, subcutaneously, once weekly on Days 1, 8, 15 and 22 during Cycles 1 and 2, then once every 2 weeks during Cycles 3 through 6, further once every 4 weeks, until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg: Participants received TAK-981 90 mg, infusion, intravenously, in combination with mezagitamab 600 mg, injection, subcutaneously, once weekly on Days 1, 8, 15, 22 during Cycles 1 and 2, then every 2 weeks during Cycles 3 through 6, further once every 4 weeks until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg | Total
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (19.29) | 65.0 (4.58) | 66.2 (12.97) | 74.0 (4.00) | 71.9 (3.94) | 68.0 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 1 | 2 | 8
  Male | 3 | 2 | 6 | 2 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 10 | 2 | 8 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 2 | 6
  White | 2 | 2 | 7 | 2 | 6 | 19
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b, Part 1: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were adverse events (AEs) that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. Adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 13 months)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
Participants | 3 | 3 | 10 | 3 | 8

2. Primary Outcome: Phase 1b, Part 1: Number of Participants With Grade 3 or Higher TEAEs
Description: The severity grade was evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0, except for Cytokine Release Syndrome (CRS), which was assessed by American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading. Where Grade 3 was severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL), Grade 4 was 4 Life-threatening consequences; urgent intervention indicated. and Grade 5 was death related to AE. TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 13 months)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
Participants | 0 | 3 | 7 | 3 | 7

3. Primary Outcome: Phase 1b, Part 1: Number of Participants With Dose Limiting Toxicities (DLTs) Based on NCI CTCAE Version 5.0
Description: DLTs were evaluated according to NCI CTCAE version 5.0. Grade 5 AE. Hematologic toxicity: Nonfebrile Grade 4 neutropenia/Grade greater than or equal to (>=) 3 febrile neutropenia; Significant Grade 3 thrombocytopenia; Grade 4 anemia or thrombocytopenia. Nonhematologic Grade 3 or higher toxicities; Grade 2 nonhematologic toxicities leading to dose reduction/discontinuation. Delay in Cycle 2 by greater than (>) 14 days or missed >1 planned doses of TAK-981/monoclonal antibody (mAb) in Cycle 1 due to TEAEs.
Time Frame: Cycle 1 (Cycle length = 28 Days)
Population: DLT-evaluable analysis set included participants who received at least 75 precent (%) of planned TAK-981 doses, all mAb doses, and have completed Cycle 1 procedures, or experienced a DLT in Cycle 1 in the phase 1 portion of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 7
Participants | 0 | 0 | 1 | 1 | 1

4. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR: percentage of participants who achieve complete response (CR) or partial response (PR) or better per investigator assessment by IMWG.CR: Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5 percent (%) plasma cells in bone marrow (BM). PR: >50 percent (%) reduction of serum M-protein and reduction in 24 hours (h) urinary M-protein by >90% or to less than (<) 200 milligrams per 24 hour (mg/24 h); If serum and urine M-protein were unmeasurable, >50% decrease in difference between involved and uninvolved free light chain (FLC) levels was required in place of M-protein criteria; If serum and urine M-protein are not measurable, and serum free light assay was also not measurable, >50% reduction in plasma cells is required in place of M-protein, provided baseline BM plasma cell percentage was >30%. In addition to the above listed criteria, if present at baseline, a >50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From date of treatment start to until date of first PD or death (whichever occurred first), up to 24 months
Population: The study was terminated after completion of Phase 1b Part 1, therefore, no participants were enrolled in Phase 2 part of the study. Hence, the data for this outcome measure could not collected, analyzed and reported.
Groups:
- Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody: Participants were planned to receive TAK-981 recommended phase 2 dose (RP2D), infusion, intravenously, in combination with an anti-CD38 antibody (mezagitamab or daratumumab and hyaluronidase-fihj), injection, subcutaneously, for up to 24 cycles or until disease progression or unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first. Each Cycle length was 28 days.
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 1b, Part 1: Observed Plasma Concentration of TAK-981
Description: Observed plasma concentration of TAK-981 was reported.
Time Frame: Cycle 1 Day 1: Pre-dose, at end of infusion (EOI), 2, 4, 6, and 24 hours post-dose; Cycle 1 Days 8 and 15: Pre-dose and EOI; Cycle 2 Days 1 and 15: Pre-dose and EOI (Cycle length = 28 days)
Population: Pharmacokinetic (PK) analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "number analyzed" signifies participants evaluable at specified time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: Predose | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ).
  Cycle 1 Day 1: EOI: number analyzed (Participants) | 2 | 1 | 9 | 1 | 6
  Cycle 1 Day 1: EOI | 225 (44.3) | 642 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 617 (61.7) | 1120 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 842 (27.5)
  Cycle 1 Day 1: 2 hours: number analyzed (Participants) | 3 | 3 | 10 | 3 | 7
  Cycle 1 Day 1: 2 hours | 79.4 (51.7) | 110 (27.8) | 115 (49.3) | 139 (47.9) | 116 (38.3)
  Cycle 1 Day 1: 4 hours: number analyzed (Participants) | 3 | 3 | 10 | 3 | 7
  Cycle 1 Day 1: 4 hours | 37.5 (45.7) | 63.0 (37.3) | 69.6 (62.3) | 63.2 (18.9) | 56.5 (38.9)
  Cycle 1 Day 1: 6 hours: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0
  Cycle 1 Day 1: 6 hours | 31.0 (65.4) | 33.2 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. |  |  |
  Cycle 1 Day 1: 24 hours: number analyzed (Participants) | 3 | 3 | 9 | 3 | 7
  Cycle 1 Day 1: 24 hours | 3.27 (68.3) | 5.91 (12.9) | 4.75 (54.0) | 5.51 (41.2) | 6.29 (57.7)
  Cycle 1 Day 8: Predose: number analyzed (Participants) | 3 | 3 | 10 | 3 | 7
  Cycle 1 Day 8: Predose | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | 0.519 (62.6) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | 0.411 (78.8) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ).
  Cycle 1 Day 8: EOI: number analyzed (Participants) | 2 | 2 | 6 | 2 | 7
  Cycle 1 Day 8: EOI | 318 (84.6) | 576 (17.1) | 829 (52.7) | 1360 (41.1) | 1070 (45.4)
  Cycle 1 Day 15: Predose: number analyzed (Participants) | 3 | 3 | 8 | 2 | 6
  Cycle 1 Day 15: Predose | 0.177 (28.8) | 0.758 (1139.8) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ).
  Cycle 1 Day 15: EOI: number analyzed (Participants) | 3 | 3 | 6 | 1 | 5
  Cycle 1 Day 15: EOI | 281 (38.1) | 585 (41.8) | 812 (55.5) | 830 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 940 (24.6)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 2 | 3 | 5 | 2 | 6
  Cycle 2 Day 1: Predose | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ).
  Cycle 2 Day 1: EOI: number analyzed (Participants) | 2 | 3 | 5 | 1 | 3
  Cycle 2 Day 1: EOI | 212 (13.1) | 844 (38.5) | 767 (61.6) | 1580 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 820 (8.7)
  Cycle 2 Day 15: Predose: number analyzed (Participants) | 2 | 1 | 3 | 1 | 5
  Cycle 2 Day 15: Predose | 0.182 (34.9) | 0.536 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | 0.286 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ).
  Cycle 2 Day 15: EOI: number analyzed (Participants) | 1 | 0 | 2 | 1 | 4
  Cycle 2 Day 15: EOI | 191 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. |  | 634 (46.3) | 1500 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 713 (14.2)

6. Secondary Outcome: Phase 1b, Part 1, Cmax: Maximum Observed Plasma Concentration for TAK-981
Description: Cmax for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: PK analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 9 | 1 | 6
ng/mL | 225 (44.3) | 642 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 617 (61.7) | 1120 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 842 (27.5)

7. Secondary Outcome: Phase 1b, Part 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-981
Description: Tmax for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 9 | 1 | 5
hours | 0.97 [0.92 to 1.02] | 1.12 [1.12 to 1.12] | 1.09 [1.00 to 1.25] | 1.09 [1.09 to 1.09] | 1.15 [1.09 to 1.25]

8. Secondary Outcome: Phase 1b, Part 1, AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for TAK-981
Description: AUC0-t for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 8 | 1 | 5
hours*nanogram per milliliter (h*ng/mL) | 813 (30.4) | 1550 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 1590 (33.9) | 2120 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 1690 (19.8)

9. Secondary Outcome: Phase 1b, Part 1, AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-981
Description: AUC0-inf for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 7 | 1 | 4
h*ng/mL | 839 (32.5) | 1590 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 1590 (36.1) | 2180 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 1690 (22.2)

10. Secondary Outcome: Phase 1b, Part 1, t1/2z: Terminal Disposition Phase Half-life for TAK-981
Description: t1/2z for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 7 | 1 | 4
hours | 5.24 [4.84 to 5.65] | 5.25 [5.25 to 5.25] | 4.96 [4.75 to 6.23] | 5.33 [5.33 to 5.33] | 5.49 [5.09 to 5.84]

11. Secondary Outcome: Phase 1b, Part 1, CL: Total Clearance for TAK-981
Description: CL for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 7 | 1 | 4
liters per hour (L/h) | 71.5 (32.5) | 56.5 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 56.7 (36.1) | 55.0 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 71.2 (22.2)

12. Secondary Outcome: Phase 1b, Part 1, Vss: Volume of Distribution at Steady State for TAK-981
Description: Vss for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 2 | 1 | 7 | 1 | 4
liters | 377 (5.1) | 281 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 250 (49.0) | 259 (NA) — Geometric Coefficient of Variation could not be estimated due to insufficient number of participants available for analysis. | 331 (20.4)

13. Secondary Outcome: Phase 1b, Part 1: Number of Participants With Positive Anti-drug Antibodies (ADA) for TAK-981 + Mezagitamab and >= 5-fold in ADA Titer
Description: ADA positive was defined as participants who had confirmed positive ADA status in at least 1 post-baseline assessments. >=5-fold in ADA titer was defined as increase in the ADA titer value post-baseline of at least 5-fold from the positive ADA titer value at baseline.
Time Frame: Baseline up to 12 months
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
Participants
  Participants with Positive ADA | 0 | 0 | 2 | 0 | 0
  Participants with >=5-fold in ADA titer | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Phase 1b, Part 1: Serum Concentration of Mezagitamab
Description: Observed serum concentrations of mezagitumab was reported.
Time Frame: Cycles 1, 2, 3, 4, 6, 7 and 12: Day 1 pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 28 days)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug. Here "number analyzed" signifies participants evaluable at specified time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
ng/mL
  Cycle 1 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below lower limit of quantification (LLOQ).
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 4 | 2 | 6
  Cycle 2 Day 1 | 99400 (38.1) | 103000 (50.9) | 81800 (53.3) | 64900 (59.4) | 29000 (6634.0)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 1 | 4
  Cycle 3 Day 1 | 95500 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 200000 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 68400 (337.7) | 146000 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 154000 (94.7)
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Cycle 4 Day 1 | 94500 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. |  |  |  |
  Cycle 6 Day 1: number analyzed (Participants) | 2 | 1 | 1 | 0 | 1
  Cycle 6 Day 1 | 38400 (83.9) | 27000 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. | 101000 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. |  | 117000 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants.
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Cycle 7 Day 1 | 71900 (NA) — Geometric Coefficient of Variation could not be calculated due to insufficient number of participants. |  |  |  |
  Cycle 12 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  Cycle 12 Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation could not be calculated because the values were below LLOQ. |  |  |  |

15. Secondary Outcome: Phase 1b, Part 1: ORR Based on International Myeloma Working Group (IMWG) Criteria
Description: ORR: percentage of participants who achieve complete response (CR) or partial response (PR) or better per investigator assessment by IMWG.CR: Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow (BM). PR: >50 percent (%) reduction of serum M-protein and reduction in 24 hours (h) urinary M-protein by >90% or to less than (<) 200 milligrams per 24 hour (mg/24 h); If the serum and urine M-protein were unmeasurable, >50% decrease in the difference between involved and uninvolved free light chain (FLC) levels was required in place of M-protein criteria; If serum and urine M-protein are not measurable, and serum free light assay was also not measurable, >50% reduction in plasma cells is required in place of M-protein, provided baseline BM plasma cell percentage was >30%. In addition to the above listed criteria, if present at baseline, a >50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From the first dose of study drug until first disease progression (PD) or death, whichever occurred first (up to 12 months)
Population: Response-evaluable analysis set included participants with measurable disease at baseline and at least 1 posttreatment evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 6
percentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 70.8] | 16.7 [0.4 to 64.1]

16. Secondary Outcome: Phases 1b, Part 1: Clinical Benefit Rate (CBR) Based on IMWG Criteria
Description: CBR: % of participants with response of at least stable disease (SD) for >=3 months or better (stringent CR [sCR], immunophenotypic CR [iCR], molecular CR [mCR], CR, very good partial response [VGPR], PR, minimal response [MR] or SD) per investigator assessment by IMWG. sCR: CR plus normal FLC ratio, absence of clonal cells in BM. iCR: sCR plus absence of phenotypical aberrant plasma in BM with minimum of 1 million total BM cells. mCR: CR plus negative allele-specific oligonucleotide polymerase chain reaction. CR: Negative immunofixation on serum, urine, disappearance soft tissue plasmacytomas, <5% plasma cells in BM. VGPR: Serum, urine M-protein detectable by immunofixation but not on electrophoresis or >90% reduction in serum M-protein+urine M-protein level <100mg/24h. PR: >50% reduction of serum M-protein and in 24h urinary M-protein by >90% or to <200mg/24h. MR: >=25% but <=49% reduction in serum M-protein, reduction in 24h urine M-protein by 50 to 89%. SD: No CR, VGPR, PR or PD.
Time Frame: From first dose of study drug until PD or death, whichever occurred first (up to 12 months)
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 6
percentage of participants | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 11.1 [0.3 to 48.2] | 0.0 [0.0 to 70.8] | 33.3 [4.3 to 77.7]

17. Secondary Outcome: Phase 1b, Part 1: Duration of Response (DOR) Based on IMWG Criteria
Description: DOR was defined as a time from date of first documentation of a PR or better to the date of first documentation of PD based on IMWG criteria. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in BM. PR: >50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to <200 mg/24 h; If the serum and urine M-protein were unmeasurable, a >50% decrease in the difference between involved and uninvolved FLC levels was required in place of the M-protein criteria; If serum and urine M-protein are not measurable, and serum free light assay was also not measurable, >50% reduction in plasma cells is required in place of M-protein, provided baseline BM plasma cell percentage was >30%. In addition to the above listed criteria, if present at baseline, a >50% reduction in the size of soft tissue plasmacytomas is also required. DOR was calculated for those participants with a confirmed PR or CR.
Time Frame: From first documented confirmed CR or PR until first documentation of PD or death, whichever occurred first (up to 12 months)
Population: Response-evaluable analysis set included participants with measurable disease at baseline and at least 1 posttreatment evaluation. Here, 'overall number of participants analyzed' signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
months |  |  |  |  | 3.2 [NA to NA] — Upper and lower limit of 95% confidence internal (CI) could not be estimated due to insufficient events.

18. Secondary Outcome: Phases 1b, Part 1: Time to Progression (TTP) Based on IMWG Criteria
Description: TTP: time from date of first dose to date of first documentation of PD as defined by standard disease criteria. PD was defined as increase of >25% from lowest response value in any one or more of following: a) Serum M-component and/or (the absolute increase must be >0.5 grams per deciliter [g/dL]). b) Urine M-component and/or (the absolute increase must be >200 mg/24 h). c) Only in participants without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be >10 milligrams per deciliter (mg/dL). d) Bone marrow plasma cell percentage; the absolute percentage must be >10%. e) Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas. f) Development of hypercalcaemia (corrected serum calcium >11.5 mg/dL or 2.65 millimoles per liter [mmol/L]) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: From first dose of study drug to the date of the first documentation of PD or death, whichever occurred first (up to 12 months)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
months | 7.9 [5.7 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 1.0 [1.0 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 1.2 [1.0 to 2.7] | 1.6 [1.2 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 3.7 [2.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events.

19. Secondary Outcome: Phases 1b, Part 1: Time to Next Treatment (TTNT)
Description: TTNT was defined as the time from the date of first dose to the date of the first dose initiation of the next line of antineoplastic therapy, for any reason.
Time Frame: From the date of first dose of study drug to the date of the first dose initiation of the next line of antineoplastic therapy (up to 12 months)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
months | 10.6 [8.6 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 5.2 [2.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 1.6 [1.5 to 6.2] | NA [2.1 to NA] — Median and Upper limit of 95% CI could not be estimated due to insufficient events. | 6.3 [1.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events.

20. Secondary Outcome: Phases 1b, Part 1: Progression-free Survival (PFS) Based on IMWG Criteria
Description: PFS was defined as time from the date of the first dose administration to the date of first documentation of PD or death due to any cause whichever occurs first. PD was defined as increase of >25% from lowest response value in any one or more of the following: a) Serum M-component and/or (the absolute increase must be >0.5 g/dL). b) Urine M-component and/or (the absolute increase must be >200 mg/24h). c) Only in participants without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dL. d) Bone marrow plasma cell percentage; the absolute percentage must be >10%. e) Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas. f) Development of hypercalcaemia (corrected serum calcium >11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: From the first dose of study drug to date of PD or death, whichever occurred first (up to 12 months)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
months | 7.9 [5.7 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 1.0 [1.0 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 1.2 [1.0 to 2.7] | 1.6 [1.2 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 3.7 [2.4 to 5.6]

21. Secondary Outcome: Phases 1b, Part 1: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death. OS was analyzed using Kaplan-Meier (KM) method. Participants were followed for survival after the last dose of study drug.
Time Frame: From date of first dose of study drug up to death from any cause (up to 27 months)
Population: Safety analysis set included participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 3 | 10 | 3 | 8
months | NA [NA to NA] — Median and upper and lower limit of 95% CI could not be estimated due to insufficient events. | NA [7.2 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient events. | 13.8 [10.9 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | 10.3 [NA to NA] — Upper limit and lower limit of 95% CI could not be estimated due to insufficient events. | 11.0 [6.5 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events.

22. Secondary Outcome: Phases 1b, Part 1: Fold Change From Baseline in Level of TAK-981-Small Ubiquitin-like Modifier (TAK-981-SUMO) Adduct Formation in Peripheral Blood Lymphocytes
Description: Blood samples were collected to assess TAK-981-SUMO adduct formation. TAK-981-SUMO adduct formation in peripheral blood lymphocytes was tested by flow cytometry with an antibody recognizing the TAK-981-SUMO adduct formation during the inhibition of the SUMO-activating enzyme by TAK-981.
Time Frame: Cycle 1 Day 1: 1, 4, and 24 hours post-dose; Cycle 1 Day 8: Pre-dose, and 1 hour post-dose; Cycle 1 Day 15: Pre-dose (Cycle length = 28 days)
Population: Pharmacodynamic analysis set included participants who provided evaluable blood samples (Cycle 1 Day 1 predose sample and at least 1 postdose sample). Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and here, "number analyzed" signifies participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 2 | 6 | 2 | 5
fold change
  Cycle 1 Day 1: 1 hour post-dose | 4.3 (0.81) | 5.1 (1.00) | 3.9 (2.63) | 5.7 (2.11) | 6.1 (4.14)
  Cycle 1 Day 1: 4 hour post-dose: number analyzed (Participants) | 0 | 1 | 5 | 2 | 4
  Cycle 1 Day 1: 4 hour post-dose |  | 4.3 (NA) — Standard Deviation could not be estimated due to insufficient number of participants available for analysis. | 3.7 (1.47) | 4.0 (0.14) | 4.1 (1.06)
  Cycle 1 Day 1: 24 hour post-dose: number analyzed (Participants) | 3 | 2 | 4 | 1 | 5
  Cycle 1 Day 1: 24 hour post-dose | 2.4 (1.12) | 3.8 (0.65) | 2.2 (0.62) | 3.5 (NA) — Standard Deviation could not be estimated due to insufficient number of participants available for analysis. | 4.4 (1.60)
  Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 2 | 2 | 5 | 2 | 3
  Cycle 1 Day 8: Pre-dose | 1.6 (0.01) | 2.5 (0.30) | 1.8 (0.78) | 2.4 (0.07) | 2.2 (0.39)
  Cycle 1 Day 8: 1 hour post-dose: number analyzed (Participants) | 2 | 2 | 6 | 2 | 3
  Cycle 1 Day 8: 1 hour post-dose | 3.5 (0.03) | 4.0 (1.18) | 6.0 (2.83) | 4.1 (0.35) | 5.6 (1.12)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 0 | 0 | 4 | 1 | 4
  Cycle 1 Day 15: Pre-dose |  |  | 1.4 (0.61) | 2.8 (NA) — Standard Deviation could not be estimated due to insufficient number of participants available for analysis. | 2.3 (0.89)

23. Secondary Outcome: Phases 1b, Part 1: Fold Change From Baseline in SUMO Pathway Inhibition in Peripheral Blood Lymphocytes
Description: Blood samples were collected to assess SUMO inhibition. SUMO pathway inhibition in peripheral blood lymphocytes was tested by flow cytometry with an antibody recognizing SUMO-2/3 chains.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
Number analyzed (Participants) | 3 | 2 | 6 | 2 | 6
fold change
  Cycle 1 Day 1: 1 hour post-dose | 0.8 (0.14) | 0.5 (0.08) | 0.7 (0.30) | 0.5 (0.16) | 1.3 (1.51)
  Cycle 1 Day 1: 4 hour post-dose: number analyzed (Participants) | 0 | 1 | 5 | 2 | 4
  Cycle 1 Day 1: 4 hour post-dose |  | 0.6 (NA) — Standard deviation could not be estimated due to insufficient number of participants available for analysis. | 0.6 (0.29) | 0.9 (0.03) | 0.7 (0.30)
  Cycle 1 Day 1: 24 hour post-dose: number analyzed (Participants) | 3 | 2 | 4 | 1 | 5
  Cycle 1 Day 1: 24 hour post-dose | 0.7 (0.08) | 0.6 (0.01) | 0.7 (0.20) | 0.8 (NA) — Standard deviation could not be estimated due to insufficient number of participants available for analysis. | 1.6 (1.85)
  Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 2 | 2 | 5 | 2 | 4
  Cycle 1 Day 8: Pre-dose | 0.6 (0.42) | 0.6 (0.24) | 0.8 (0.23) | 0.6 (0.58) | 1.5 (1.09)
  Cycle 1 Day 8: 1 hour post-dose: number analyzed (Participants) | 2 | 2 | 6 | 2 | 4
  Cycle 1 Day 8: 1 hour post-dose | 0.4 (0.25) | 0.3 (0.19) | 0.6 (0.61) | 0.4 (0.29) | 1.3 (1.56)
  Cycle 1 Day 15: Pre-dose: number analyzed (Participants) | 0 | 0 | 4 | 1 | 5
  Cycle 1 Day 15: Pre-dose |  |  | 0.5 (0.39) | 0.8 (NA) — Standard deviation could not be estimated due to insufficient number of participants available for analysis. | 4.0 (5.38)

24. Secondary Outcome: Phase 2: Number of Participants With TEAEs and TEAEs by Severity
Description: TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product. The severity grade was evaluated as per the NCI CTCAE Version 5.0, except for CRS, which was assessed by ASTCT consensus grading. Where Grade 3 was severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4 was 4 Life-threatening consequences; urgent intervention indicated. and Grade 5 was death related to AE. TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug.
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

25. Secondary Outcome: Phase 2: CBR Based on IMWG Criteria
Description: CBR: percentage of participants with response of at least (SD for >=3 months or better sCR, iCR, mCR, CR, very good partial response [VGPR], PR, minimal response [MR] or SD) per investigator assessment by IMWG. sCR: CR plus normal FLC ratio, absence of clonal cells in BM. iCR: sCR plus absence of phenotypical aberrant plasma in BM with minimum of 1 million total BM cells. mCR: CR plus negative allele-specific oligonucleotide polymerase chain reaction. CR: Negative immunofixation on serum, urine, disappearance soft tissue plasmacytomas, <5% plasma cells in BM. VGPR: Serum, urine M-protein detectable by immunofixation but not on electrophoresis or >90% reduction in serum M-protein+urine M-protein level <100mg/24h. PR: >50% reduction of serum M-protein and in 24h urinary M-protein by >90% or to <200mg/24h. MR:>=25% but <=49% reduction in serum M-protein, reduction in 24h urine M-protein by 50 to 89%. SD: No CR, VGPR, PR or PD.
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

26. Secondary Outcome: Phase 2: DOR Based on IMWG Criteria
Description: DOR was defined as a time from date of first documentation of a PR or better to the date of first documentation of PD based on IMWG criteria. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in BM. PR: >50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to <200 mg/24 h; If the serum and urine M-protein were unmeasurable, a >50% decrease in the difference between involved and uninvolved FLC levels was required in place of the M-protein criteria; If serum and urine M-protein are not measurable, and serum free light assay was also not measurable, >50% reduction in plasma cells is required in place of M-protein, provided baseline BM plasma cell percentage was >30%. In addition to the above listed criteria, if present at baseline, a >50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

27. Secondary Outcome: Phase 2: TTP Based on IMWG Criteria
Description: TTP: time from date of first dose to date of first documentation of PD as defined by standard disease criteria. PD was defined as increase of >25% from lowest response value in any one or more of following: a) Serum M-component and/or (the absolute increase must be >0.5 grams per deciliter [g/dL]). b) Urine M-component and/or (the absolute increase must be >200 mg/24 h). c) Only in participants without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be >10 milligrams per deciliter (mg/dL). d) Bone marrow plasma cell percentage; the absolute percentage must be >10%. e) Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas. f) Development of hypercalcaemia (corrected serum calcium >11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

28. Secondary Outcome: Phase 2: Time to Next Treatment (TTNT)
Description: as for outcome 19
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

29. Secondary Outcome: Phase 2: PFS Based on IMWG Criteria
Description: as for outcome 20
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

30. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death.
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

31. Secondary Outcome: Phase 2: Percentage of Participants With MRD Negative Status as Determined by Next-Generation Sequencing (NGS)
Time Frame: Up to 24 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

32. Secondary Outcome: Phase 2: Minimal Residual Disease (MRD) Negative Rate
Time Frame: Up to 12 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

33. Secondary Outcome: Phase 2: Durable MRD Negative Rate
Time Frame: Up to 12 months
Population: as for outcome 4
Arm/Group | Phase 2: TAK-981 (RP2D) + Selected Anti-CD38 Antibody
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 13 months)
Description: The study was terminated after completion of Phase 1b Part 1, therefore, no participants were enrolled in Phase 1b-Part 2 and Phase 2 of this study. Hence, no safety data for Phase 1b-Part 2 and Phase 2 was collected, analyzed and reported in this AEs section.
Arm/Group | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 4/10 | 1/3 | 4/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 4/10 | 1/3 | 3/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/10 | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg (N=3) | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg (N=3) | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg (N=10) | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg (N=3) | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg (N=8)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Part 1: TAK-981 60 mg BIW + Mezagitamab 600 mg (N=3) | Phase 1b, Part 1: TAK-981 90 mg BIW + Mezagitamab 600 mg (N=3) | Phase 1b, Part 1: TAK-981 90 mg QW + Mezagitamab 600 mg (N=10) | Phase 1b, Part 1: TAK-981 120 mg BIW + Mezagitamab 600 mg (N=3) | Phase 1b, Part 1: TAK-981 120 mg QW + Mezagitamab 600 mg (N=8)
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0 | 2
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 3
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 5
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Epidural lipomatosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 4 | 2 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 2 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Platelet count decreased (Investigations) | 1 | 1 | 1 | 3 | 2
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 2
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 1 | 1
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT04776018/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT04776018/SAP_001.pdf